CLINICAL TRIAL: NCT06738355
Title: PREVENT: Practice-based Approaches to Promote HPV Vaccination in the Safety Net - Pilot Trial
Brief Title: PREVENT Pilot HPV - Related Cancers Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Utah (Other)
Collaborators: Kaiser Permanente (Other); University of Arizona (Other); Sea Mar Community Health Centers (Other); National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Prevention
Other Study IDs: HCI161649-2; 1R01CA279973-01 (NIH); DSS_10065815 (Other: University of Utah, Document Summary Sheet (DSS) Number)
Record Dates: First submitted 2024-12-12; First posted 2024-12-17 (Actual); Last update posted 2025-09-24 (Actual); Status verified 2025-09

CONDITIONS: HPV Vaccination; Uptake Vaccination; Series Completion
Keywords: Humans; Adolescent; Child; Male; Female; Caregivers; Parents; Hispanic or Latino; Rural Population; Health Personnel; United States; Vaccination; Papillomavirus Vaccines; Papillomavirus Vaccines / administration & dosage; Human Papillomavirus Viruses; Papillomavirus Infections; Papillomavirus Infections / prevention & control; Cancer / prevention & control; Incidence; Text Messaging; Reminder Systems / instrumentation; Social Norms; Vaccination Refusal; Health Knowledge, Attitudes, Practice; Health Promotion / methods; Motivation; Communication; Patient Acceptance of Health Care; Parents / education; Religion; Religiosity; Stakeholder Participation; Participatory Approach; Qualitative Research; Quantitative Research; Randomized Control Trial; Surveys and Questionnaires
MeSH Terms: conditions — Papillomavirus Infections; Neoplasms; Vaccination Refusal; Behavior; Communication; Patient Acceptance of Health Care

STUDY DESIGN:
Intervention Model Description: The investigators will use intervention mapping (IM) to plan each intervention step. The investigators will apply IM to develop and test HPV vaccination reminders for parents/caregivers (P/C).
  Intervention: The investigators propose a 3-arm pilot trial to assess the feasibility of a RCT comparing rates of completing the next step in the HPV vaccination series at six months and completing the HPV vaccination series at 13 months between Auto, Auto-Plus, and UC arms. P/C of children/adolescents (C/A) who have not completed the series will be randomized 1:1:1 to study arms. Participants will be assessed for eligibility and enrolled, with a total participant time in the study of 13 months, for a total of 25 months of enrollment, participation, and follow-up.
Who Masked: Participant, Care Provider
Masking Description: Clinic analysts will create a real-time list of patients due for an initial HPV vaccine dose. P/C of remaining C/A patients will be individually randomized to either Auto or Auto-Plus intervention or usual care (UC) in a 1:1:1 ratio. This study will only target one child/adolescent per parent/caregiver (siblings will be excluded from intervention assessments). The investigators will select a cohort of 519 P/C patients from the 4 clinics, randomized to intervention arms (UC, Auto, and Auto-Plus). Intervention activities largely mimic clinic processes, and clinicians and participants will be unaware of which intervention study arm the P/C has been assigned.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Automated Intervention (Auto) (Experimental): Auto intervention participants will be eligible for outreach delivered using automated phone calls, text, or email messages with the mode, frequency, timing of reminders, and message content. Automated outreach may also include innovative communication strategies, such as text-linked videos, P/C, or patient narratives. Auto outreach to P/C will invite P/Cs to attend free HPV vaccination visits and emphasize family-friendly hours.
  Interventions: Behavioral: PREVENT
- Automated Intervention Plus (Auto-Plus) (Experimental): Auto-Plus intervention participants will be eligible for automated reminders, plus additional P/C prompts for patients who do not undergo vaccination within three weeks. These prompts may be delivered via live phone call outreach or patient navigation. Activities selected from a list of possible options from the National HPV Vaccination Roundtable and our ranking of the effectiveness of language- and culturally-tailored intervention materials.
  Interventions: Behavioral: PREVENT
- Usual Care (UC) (No Intervention): The UC group will not receive tailored reminders but will only receive opportunistic vaccine reminders that are delivered during clinic visits or MyChart EHR-based patient portal reminders.

INTERVENTIONS:
Behavioral: PREVENT — The proposed study will assess the feasibility of an RCT for clinic-based outreach to increase vaccination rates for HPV at community clinics in rural counties. The study is a pilot trial that will assign adult parent/caregiver participants to a timeline for receiving the vaccination messaging intervention. Auto and Auto-Plus intervention arms may use some of the same components (automated calls, live calls, text messages, emails, and mailings).
  Arms: Automated Intervention (Auto); Automated Intervention Plus (Auto-Plus)

SUMMARY:
This study will serve as one of the first to develop and test the effectiveness of strategies to promote HPV vaccination among diverse rural parents and caregivers of children ages 9-17 years in the Mountain West. Once implemented into practice, our intervention could significantly reduce disparities in the burden of HPV-associated cancers among rural populations in the United States.

The proposed study will assess the feasibility of clinic-based outreach to increase vaccination rates for HPV at four community clinics in rural counties in Washington.

DETAILED DESCRIPTION:
This is a randomized, pilot study two human papillomavirus (HPV) vaccination patient reminder intervention arms that will take place in rural clinics operated by Sea Mar Community Health Centers.

The PREVENT PILOT study will administer a three-arm, patient-randomized controlled trial that will assess the feasibility of clinic-based outreach to increase vaccination rates. The study arms will consist of automated reminders, automated plus live reminders, and usual care. Parents/caregivers of children and adolescents selected for the trial will be chosen using established study criteria applied to the electronic health records linked to state immunization registries. As a minimal-risk study, for the intervention only, the investigators will apply for a waiver of informed consent. The PILOT study will be delivered as part of standard care, and patients will be unaware they are in the trial. Delivered vaccination messages will include opt-out choices.

Parents/caregivers (P/C) of children and adolescents (C/A) will be sent any number of reminders to encourage parents to obtain an HPV vaccine for their age-eligible C/A. Reminders may include text messages, automated phone calls, mailed letters, live calls, or patient navigation. Reminders will be delivered by a vendor (automated reminders) or clinic staff (live reminders). Reminders will be delivered in English and Spanish, and interpreter services may be used for live reminders to the small proportion of patients who speak languages other than English or Spanish.

The primary objective of this pilot study is the feasibility of the trial, which will be assessed by the number of patients randomized to the study intervention. Other secondary outcome measures include the correctness of the randomization, successful receipt of a text message intervention, the proportion of participants who responded to the text intervention, and the proportion of participants who were successfully contacted.

During active study recruitment, the investigators will convene a meeting of our data safety monitor board every six months. The investigators will disseminate study findings and research products in accordance with our dissemination plan. The study findings will serve as a basis for a larger multi-level trial of HPV vaccination in rural communities.

ELIGIBILITY:
Inclusion Criteria:

1. Parents/Caregivers (P/C) of children/adolescents (C/A) ages 9-17 years of age (i.e., age-eligible for HPV vaccination);
2. P/C with active clinic patients (i.e., have been seen in the clinic in the last 12 months); and
3. P/C who speak either English or Spanish.

Exclusion Criteria:

1. P/C of C/A with previous excluding HPV vaccination history (e.g., completed vaccination, or not due);
2. P/C of C/A with clinical conditions that influence the CDC HPV vaccination recommendations (e.g., pregnancy);
3. P/C of C/A with other factors that would influence CDC HPV recommendations; and
4. P/C that does not speak Spanish or English.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 519 (Actual)
Dates: Start 2025-05-20 (Actual); Primary Completion 2025-08-12 (Actual); Study Completion 2025-08-12 (Actual)

PRIMARY OUTCOMES:
Number of Participants Correctly Randomized | up to 1 day after randomization
  To assess the feasibility of the study intervention. This outcome measure will report the count of participants who were correctly randomized according to the study protocol.

SECONDARY OUTCOMES:
Number of Participants Who Responded to the Text Intervention | up to 1 month after randomization
  To assess the feasibility of the study intervention. This outcome measure will report the number of participants who responded to the text-based intervention, as defined by the study protocol.
Proportion of Participants Successfully Contacted | up to 1 day
  To assess the feasibility of the study intervention. This outcome measure will report the proportion of participants who were successfully contacted out of the total number of attempted contacts.

CONTACTS AND LOCATIONS:
Overall Officials: Deanna Kepka, PhD, MPH, Principal Investigator — Study Principal Investigator
Locations (1):
- Sea Mar Community Health Centers, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: Undecided
A plan for sharing IDP that maintains participant anonymity has not yet been developed.

REFERENCES:
- [Background] Saslow D, Andrews KS, Manassaram-Baptiste D, Loomer L, Lam KE, Fisher-Borne M, Smith RA, Fontham ET; American Cancer Society Guideline Development Group. Human papillomavirus vaccination guideline update: American Cancer Society guideline endorsement. CA Cancer J Clin. 2016 Sep;66(5):375-85. doi: 10.3322/caac.21355. Epub 2016 Jul 19. PMID 27434803
- [Background] Tabak RG, Duggan K, Smith C, Aisaka K, Moreland-Russell S, Brownson RC. Assessing Capacity for Sustainability of Effective Programs and Policies in Local Health Departments. J Public Health Manag Pract. 2016 Mar-Apr;22(2):129-37. doi: 10.1097/PHH.0000000000000254. PMID 25946700
- [Background] Brownson RC, Reis RS, Allen P, Duggan K, Fields R, Stamatakis KA, Erwin PC. Understanding administrative evidence-based practices: findings from a survey of local health department leaders. Am J Prev Med. 2014 Jan;46(1):49-57. doi: 10.1016/j.amepre.2013.08.013. PMID 24355671
- [Background] Shea CM, Jacobs SR, Esserman DA, Bruce K, Weiner BJ. Organizational readiness for implementing change: a psychometric assessment of a new measure. Implement Sci. 2014 Jan 10;9:7. doi: 10.1186/1748-5908-9-7. PMID 24410955
- [Background] Wutich A, Bernard HR. Sharing qualitative data & analysis. With whom and how widely?: A response to 'Promises and pitfalls of data sharing in qualitative research'. Soc Sci Med. 2016 Nov;169:199-200. doi: 10.1016/j.socscimed.2016.09.041. Epub 2016 Sep 30. No abstract available. PMID 27720554
- [Background] Patton MQ. Qualitative research and evaluation methods. Thousand Oaks, CA: Sage Publications, Inc.; 2002
- [Background] Malterud K, Siersma VD, Guassora AD. Sample Size in Qualitative Interview Studies: Guided by Information Power. Qual Health Res. 2016 Nov;26(13):1753-1760. doi: 10.1177/1049732315617444. Epub 2016 Jul 10. PMID 26613970
- [Background] Silverman D. Qualitative Research: A practical handbook. Thousand Oaks, CA: Sage Publications, Inc.; 2010.
- [Background] Nonzee NJ, Baldwin SB, Cui Y, Singhal R. Disparities in parental human papillomavirus (HPV) vaccine awareness and uptake among adolescents. Vaccine. 2018 Feb 28;36(10):1243-1247. doi: 10.1016/j.vaccine.2017.08.046. Epub 2017 Sep 28. PMID 28967520
- [Background] Choi Y, Eworuke E, Segal R. What explains the different rates of human papillomavirus vaccination among adolescent males and females in the United States? Papillomavirus Res. 2016 Dec;2:46-51. doi: 10.1016/j.pvr.2016.02.001. Epub 2016 Mar 4. PMID 29074185
- [Background] Warner EL, Ding Q, Pappas L, Bodson J, Fowler B, Mooney R, Kirchhoff AC, Kepka D. Health Care Providers' Knowledge of HPV Vaccination, Barriers, and Strategies in a State With Low HPV Vaccine Receipt: Mixed-Methods Study. JMIR Cancer. 2017 Aug 11;3(2):e12. doi: 10.2196/cancer.7345. PMID 28801303
- [Background] Garcia AA, Zuniga JA, Lagon C. A Personal Touch: The Most Important Strategy for Recruiting Latino Research Participants. J Transcult Nurs. 2017 Jul;28(4):342-347. doi: 10.1177/1043659616644958. Epub 2016 Apr 25. PMID 27114390
- [Background] Kim SY, Chen S, Hou Y, Zeiders KH, Calzada EJ. Parental socialization profiles in Mexican-origin families: Considering cultural socialization and general parenting practices. Cultur Divers Ethnic Minor Psychol. 2019 Jul;25(3):439-450. doi: 10.1037/cdp0000234. Epub 2018 Nov 1. PMID 30382707
- [Background] Coronado GD, Petrik A, Spofford M, Talbot J, Do HH, Sanchez J, Kapka T, Taylor V. Perceptions of under and overutilization of cervical cancer screening services at Latino-serving community health centers. J Community Health. 2013 Oct;38(5):915-8. doi: 10.1007/s10900-013-9701-1. PMID 23728821
- [Background] Jackson ML, Henrikson NB, Grossman DC. Evaluating Washington State's immunization information system as a research tool. Acad Pediatr. 2014 Jan-Feb;14(1):71-6. doi: 10.1016/j.acap.2013.10.002. PMID 24369871
- [Background] Maneesriwongul W, Dixon JK. Instrument translation process: a methods review. J Adv Nurs. 2004 Oct;48(2):175-86. doi: 10.1111/j.1365-2648.2004.03185.x. PMID 15369498
- [Background] Centers for Disease Control and Prevention. Human Papillomavirus (HPV). Educational Materials. Available from: https://www.cdc.gov/hpv/hcp/educational-materials.html.
- [Background] Moorhead SA, Hazlett DE, Harrison L, Carroll JK, Irwin A, Hoving C. A new dimension of health care: systematic review of the uses, benefits, and limitations of social media for health communication. J Med Internet Res. 2013 Apr 23;15(4):e85. doi: 10.2196/jmir.1933. PMID 23615206
- [Background] Pew Research Center. Mobile Fact Sheet. Available from: https://www.pewresearch.org/internet/fact-sheet/mobile/
- [Background] Tiro JA, Sanders JM, Pruitt SL, Stevens CF, Skinner CS, Bishop WP, Fuller S, Persaud D. Promoting HPV Vaccination in Safety-Net Clinics: A Randomized Trial. Pediatrics. 2015 Nov;136(5):850-9. doi: 10.1542/peds.2015-1563. Epub 2015 Oct 19. PMID 26482674
- [Background] Calo WA, Gilkey MB, Malo TL, Robichaud M, Brewer NT. A content analysis of HPV vaccination messages available online. Vaccine. 2018 Nov 26;36(49):7525-7529. doi: 10.1016/j.vaccine.2018.10.053. Epub 2018 Oct 23. PMID 30366803
- [Background] Nan X, Madden K, Richards A, Holt C, Wang MQ, Tracy K. Message Framing, Perceived Susceptibility, and Intentions to Vaccinate Children Against HPV Among African American Parents. Health Commun. 2016 Jul;31(7):798-805. doi: 10.1080/10410236.2015.1005280. Epub 2015 Dec 8. PMID 26646190
- [Background] Mroz S, Zhang X, Williams M, Conlon A, LoConte NK. Working to Increase Vaccination for Human Papillomavirus: A Survey of Wisconsin Stakeholders, 2015. Prev Chronic Dis. 2017 Sep 28;14:E85. doi: 10.5888/pcd14.160610. PMID 28957034
- [Background] Thompson JH, Davis MM, Michaels L, Rivelli JS, Castillo ML, Younger BM, Castro M, Reich SL, Coronado GD. Developing Patient-Refined Messaging for a Mailed Colorectal Cancer Screening Program in a Latino-Based Community Health Center. J Am Board Fam Med. 2019 May-Jun;32(3):307-317. doi: 10.3122/jabfm.2019.03.180026. PMID 31068395
- [Background] National Heart Lung and Blood Institute. Research dissemination and implementation (R18) grants2011 01/09/2012. Available from: http://www.nhlbi.nih.gov/funding/policies/dissemination&implementationR18.htm.
- [Background] Glasgow RE, Klesges LM, Dzewaltowski DA, Estabrooks PA, Vogt TM. Evaluating the impact of health promotion programs: using the RE-AIM framework to form summary measures for decision making involving complex issues. Health Educ Res. 2006 Oct;21(5):688-94. doi: 10.1093/her/cyl081. Epub 2006 Aug 31. PMID 16945984
- [Background] Glasgow RE, Wagner EH, Schaefer J, Mahoney LD, Reid RJ, Greene SM. Development and validation of the Patient Assessment of Chronic Illness Care (PACIC). Med Care. 2005 May;43(5):436-44. doi: 10.1097/01.mlr.0000160375.47920.8c. PMID 15838407
- [Background] Glasgow RE, Ory MG, Klesges LM, Cifuentes M, Fernald DH, Green LA. Practical and relevant self-report measures of patient health behaviors for primary care research. Ann Fam Med. 2005 Jan-Feb;3(1):73-81. doi: 10.1370/afm.261. PMID 15671195
- [Background] Glasgow RE, Klesges LM, Dzewaltowski DA, Bull SS, Estabrooks P. The future of health behavior change research: what is needed to improve translation of research into health promotion practice? Ann Behav Med. 2004 Feb;27(1):3-12. doi: 10.1207/s15324796abm2701_2. PMID 14979858
- [Background] National Cancer Institute. How do RE-AIM elements relate to planning? 2011 01/05/2012. Available from: http://cancercontrol.cancer.gov/IS/reaim/faq.html#define.
- [Background] Glasgow RE. RE-AIMing research for application: ways to improve evidence for family medicine. J Am Board Fam Med. 2006 Jan-Feb;19(1):11-9. doi: 10.3122/jabfm.19.1.11. PMID 16492000
- [Background] Thompson JH, Davis MM, Leo MC, Schneider JL, Smith DH, Petrik AF, Castillo M, Younger B, Coronado GD. Participatory Research to Advance Colon Cancer Prevention (PROMPT): Study protocol for a pragmatic trial. Contemp Clin Trials. 2018 Apr;67:11-15. doi: 10.1016/j.cct.2018.02.001. Epub 2018 Feb 9. PMID 29408304
- [Background] Westfall JM, Zittleman L, Sutter C, Emsermann CB, Staton EW, Van Vorst R, Dickinson LM; Community Advisory Council. Testing to prevent colon cancer: results from a rural community intervention. Ann Fam Med. 2013 Nov-Dec;11(6):500-7. doi: 10.1370/afm.1582. PMID 24218373
- [Background] Norman N, Bennett C, Cowart S, Felzien M, Flores M, Flores R, Haynes C, Hernandez M, Rodriquez MP, Sanchez N, Sanchez S, Winkelman K, Winkelman S, Zittleman L, Westfall JM. Boot camp translation: a method for building a community of solution. J Am Board Fam Med. 2013 May-Jun;26(3):254-63. doi: 10.3122/jabfm.2013.03.120253. PMID 23657693
- [Background] Satcher, D. (2005). Methods in community-based participatory research for health. John Wiley & Sons.
- [Background] SeaMar Community Health Centers (Clinica de la Comunidad). Report to the Community2018 02/26/2019. Available from: https://seamar.org/seamar-downloads/Annual-Report2018.pdf
- [Background] Coronado GD, Golovaty I, Longton G, Levy L, Jimenez R. Effectiveness of a clinic-based colorectal cancer screening promotion program for underserved Hispanics. Cancer. 2011 Apr 15;117(8):1745-54. doi: 10.1002/cncr.25730. Epub 2010 Nov 8. PMID 21472722
- [Background] Edwards BK, Ward E, Kohler BA, Eheman C, Zauber AG, Anderson RN, Jemal A, Schymura MJ, Lansdorp-Vogelaar I, Seeff LC, van Ballegooijen M, Goede SL, Ries LA. Annual report to the nation on the status of cancer, 1975-2006, featuring colorectal cancer trends and impact of interventions (risk factors, screening, and treatment) to reduce future rates. Cancer. 2010 Feb 1;116(3):544-73. doi: 10.1002/cncr.24760. PMID 19998273
- [Background] Parker E, Margolis LH, Eng E, Henriquez-Roldan C. Assessing the capacity of health departments to engage in community-based participatory public health. Am J Public Health. 2003 Mar;93(3):472-6. doi: 10.2105/ajph.93.3.472. PMID 12604498
- [Background] Thompson B, Coronado G, Snipes SA, Puschel K. Methodologic advances and ongoing challenges in designing community-based health promotion programs. Annu Rev Public Health. 2003;24:315-40. doi: 10.1146/annurev.publhealth.24.100901.140819. Epub 2001 Nov 6. PMID 12471272
- [Background] University of Washington. Developing and Sustaining Community Based Participatory Research Partnerships: A Skill Building Curriculum2012 04/21/2012 Available from: http://depts.washington.edu/ccph/cbpr/u1/u11.php.
- [Background] University of Washington School of Public Health and Community Medicine. Community-based research principles. Available from: http://sphcm.washington.edu/research/community.htm.
- [Background] Byrd TL, Wilson KM, Smith JL, Coronado G, Vernon SW, Fernandez-Esquer ME, Thompson B, Ortiz M, Lairson D, Fernandez ME. AMIGAS: a multicity, multicomponent cervical cancer prevention trial among Mexican American women. Cancer. 2013 Apr 1;119(7):1365-72. doi: 10.1002/cncr.27926. Epub 2012 Dec 21. PMID 23280399
- [Background] Thompson B, Carosso EA, Jhingan E, Wang L, Holte SE, Byrd TL, Benavides MC, Lopez C, Martinez-Gutierrez J, Ibarra G, Gonzalez VJ, Gonzalez NE, Duggan CR. Results of a randomized controlled trial to increase cervical cancer screening among rural Latinas. Cancer. 2017 Feb 15;123(4):666-674. doi: 10.1002/cncr.30399. Epub 2016 Oct 27. PMID 27787893
- [Background] Duggan C, Coronado G, Martinez J, Byrd TL, Carosso E, Lopez C, Benavides M, Thompson B. Cervical cancer screening and adherence to follow-up among Hispanic women study protocol: a randomized controlled trial to increase the uptake of cervical cancer screening in Hispanic women. BMC Cancer. 2012 May 6;12:170. doi: 10.1186/1471-2407-12-170. PMID 22559251
- [Background] Coronado GD, Rivelli JS, Fuoco MJ, Vollmer WM, Petrik AF, Keast E, Barker S, Topalanchik E, Jimenez R. Effect of Reminding Patients to Complete Fecal Immunochemical Testing: A Comparative Effectiveness Study of Automated and Live Approaches. J Gen Intern Med. 2018 Jan;33(1):72-78. doi: 10.1007/s11606-017-4184-x. Epub 2017 Oct 10. PMID 29019046
- [Background] Coronado GD, Burdick T, Petrik A, Kapka T, Retecki S, Green B. Using an Automated Data-driven, EHR-Embedded Program for Mailing FIT kits: Lessons from the STOP CRC Pilot Study. J Gen Pract (Los Angel). 2014 Jan 5;2:1000141. doi: 10.4172/2329-9126.1000141. PMID 25411657
- [Background] Kepka DL, Ulrich AK, Coronado GD. Low knowledge of the three-dose HPV vaccine series among mothers of rural Hispanic adolescents. J Health Care Poor Underserved. 2012 May;23(2):626-35. doi: 10.1353/hpu.2012.0040. PMID 22643612
- [Background] Kepka DL, Coronado GD, Rodriguez HP, Thompson B. Development of a radionovela to promote HPV vaccine awareness and knowledge among Latino parents. Public Health Rep. 2012 Jan-Feb;127(1):130-8. doi: 10.1177/003335491212700118. No abstract available. PMID 22298937
- [Background] Ayres S, Gee A, Kim S, Hashibe M, Praag A, Kaiser D, Chang CP, Brandt HM, Kepka D. Human Papillomavirus Vaccination Knowledge, Barriers, and Recommendations Among Healthcare Provider Groups in the Western United States. J Cancer Educ. 2022 Dec;37(6):1816-1823. doi: 10.1007/s13187-021-02047-6. Epub 2021 Jul 8. PMID 34236651
- [Background] Brandt HM, Kepka D, Kirchhoff AC, Daniel CL, Bhatt NS. Human papillomavirus (HPV) vaccination is cancer prevention for childhood cancer survivors. Cancer. 2022 Jan 15;128(2):237-239. doi: 10.1002/cncr.33920. Epub 2021 Oct 4. PMID 34606629
- [Background] Kepka D, Christini K, McGough E, Wagner A, Del Fiol G, Gibson B, Ayres S, Brandt HM, Mann S, Petrik AF, Coronado GD. Successful Multi-Level HPV Vaccination Intervention at a Rural Healthcare Center in the Era of COVID-19. Front Digit Health. 2021 Aug 19;3:719138. doi: 10.3389/fdgth.2021.719138. eCollection 2021. PMID 34713184
- [Background] Kepka D, Ding Q, Bodson J, Warner EL, Mooney K. Latino Parents' Awareness and Receipt of the HPV Vaccine for Sons and Daughters in a State with Low Three-Dose Completion. J Cancer Educ. 2015 Dec;30(4):808-12. doi: 10.1007/s13187-014-0781-0. PMID 25572463
- [Background] Warner EL, Lai D, Carbajal-Salisbury S, Garza L, Bodson J, Mooney K, Kepka D. Latino Parents' Perceptions of the HPV Vaccine for Sons and Daughters. J Community Health. 2015 Jun;40(3):387-94. doi: 10.1007/s10900-014-9949-0. PMID 25269400
- [Background] Kepka D, Warner EL, Kinney AY, Spigarelli MG, Mooney K. Low human papillomavirus (HPV) vaccine knowledge among Latino parents in Utah. J Immigr Minor Health. 2015 Feb;17(1):125-31. doi: 10.1007/s10903-014-0003-1. PMID 24609357
- [Background] Warner EL, Ding Q, Pappas LM, Henry K, Kepka D. White, affluent, educated parents are least likely to choose HPV vaccination for their children: a cross-sectional study of the National Immunization Study - teen. BMC Pediatr. 2017 Dec 1;17(1):200. doi: 10.1186/s12887-017-0953-2. PMID 29191180
- [Background] Islam JY, Gruber JF, Kepka D, Kunwar M, Smith SB, Rothholz MC, Brewer NT, Smith JS. Pharmacist insights into adolescent human papillomavirus vaccination provision in the United States. Hum Vaccin Immunother. 2019;15(7-8):1839-1850. doi: 10.1080/21645515.2018.1556077. Epub 2019 Feb 6. PMID 30550369
- [Background] Elam-Evans LD, Yankey D, Singleton JA, Sterrett N, Markowitz LE, Williams CL, Fredua B, McNamara L, Stokley S. National, Regional, State, and Selected Local Area Vaccination Coverage Among Adolescents Aged 13-17 Years - United States, 2019. MMWR Morb Mortal Wkly Rep. 2020 Aug 21;69(33):1109-1116. doi: 10.15585/mmwr.mm6933a1. PMID 32817598
- [Background] Vogelaar I, van Ballegooijen M, Schrag D, Boer R, Winawer SJ, Habbema JD, Zauber AG. How much can current interventions reduce colorectal cancer mortality in the U.S.? Mortality projections for scenarios of risk-factor modification, screening, and treatment. Cancer. 2006 Oct 1;107(7):1624-33. doi: 10.1002/cncr.22115. PMID 16933324
- [Background] Hopfer S, Garcia S, Duong HT, Russo JA, Tanjasiri SP. A Narrative Engagement Framework to Understand HPV Vaccination Among Latina and Vietnamese Women in a Planned Parenthood Setting. Health Educ Behav. 2017 Oct;44(5):738-747. doi: 10.1177/1090198117728761. Epub 2017 Aug 30. PMID 28854812
- [Background] Szilagyi PG, Humiston SG, Gallivan S, Albertin C, Sandler M, Blumkin A. Effectiveness of a citywide patient immunization navigator program on improving adolescent immunizations and preventive care visit rates. Arch Pediatr Adolesc Med. 2011 Jun;165(6):547-53. doi: 10.1001/archpediatrics.2011.73. PMID 21646588
- [Background] Vanderpool RC, Stradtman LR, Brandt HM. Policy opportunities to increase HPV vaccination in rural communities. Hum Vaccin Immunother. 2019;15(7-8):1527-1532. doi: 10.1080/21645515.2018.1553475. Epub 2019 Jan 4. PMID 30608894
- [Background] Brandt HM, Pierce JY, Crary A. Increasing HPV vaccination through policy for public health benefit. Hum Vaccin Immunother. 2016 Jun 2;12(6):1623-5. doi: 10.1080/21645515.2015.1122145. Epub 2015 Dec 15. PMID 26669416
- [Background] Khuwaja SS, Peck JL. Increasing HPV Vaccination Rates Using Text Reminders: An Integrative Review of the Literature. J Pediatr Health Care. 2022 Jul-Aug;36(4):310-320. doi: 10.1016/j.pedhc.2022.02.001. Epub 2022 Mar 11. PMID 35288016
- [Background] Francis DB, Cates JR, Wagner KPG, Zola T, Fitter JE, Coyne-Beasley T. Communication technologies to improve HPV vaccination initiation and completion: A systematic review. Patient Educ Couns. 2017 Jul;100(7):1280-1286. doi: 10.1016/j.pec.2017.02.004. Epub 2017 Feb 6. PMID 28209248
- [Background] Hou SI, Fernandez ME, Parcel GS. Development of a cervical cancer educational program for Chinese women using intervention mapping. Health Promot Pract. 2004 Jan;5(1):80-7. doi: 10.1177/1524839903257311. PMID 14965438
- [Background] Byrd TL, Wilson KM, Smith JL, Heckert A, Orians CE, Vernon SW, Fernandez-Esquer ME, Fernandez ME. Using intervention mapping as a participatory strategy: development of a cervical cancer screening intervention for Hispanic women. Health Educ Behav. 2012 Oct;39(5):603-11. doi: 10.1177/1090198111426452. Epub 2012 Mar 1. PMID 22388451
- [Background] Fernandez ME, Gonzales A, Tortolero-Luna G, Partida S, Bartholomew LK. Using intervention mapping to develop a breast and cervical cancer screening program for Hispanic farmworkers: Cultivando La Salud. Health Promot Pract. 2005 Oct;6(4):394-404. doi: 10.1177/1524839905278810. PMID 16210681
- [Background] Warner EL, Fowler B, Martel L, Kepka D. Improving HPV Vaccination Through a Diverse Multi-state Coalition. J Community Health. 2017 Oct;42(5):911-920. doi: 10.1007/s10900-017-0334-7. PMID 28393294
- [Background] Bartholomew LK, Parcel GS, Kok G. Intervention mapping: a process for developing theory- and evidence-based health education programs. Health Educ Behav. 1998 Oct;25(5):545-63. doi: 10.1177/109019819802500502. PMID 9768376
- [Background] Paskett ED, Krok-Schoen JL, Pennell ML, Tatum CM, Reiter PL, Peng J, Bernardo BM, Weier RC, Richardson MS, Katz ML. Results of a Multilevel Intervention Trial to Increase Human Papillomavirus (HPV) Vaccine Uptake among Adolescent Girls. Cancer Epidemiol Biomarkers Prev. 2016 Apr;25(4):593-602. doi: 10.1158/1055-9965.EPI-15-1243. PMID 27196093
- [Background] Fridman A, Gershon R, Gneezy A. COVID-19 and vaccine hesitancy: A longitudinal study. PLoS One. 2021 Apr 16;16(4):e0250123. doi: 10.1371/journal.pone.0250123. eCollection 2021. PMID 33861765
- [Background] Santibanez TA, Singleton JA, Santibanez SS, Wortley P, Bell BP. Socio-demographic differences in opinions about 2009 pandemic influenza A (H1N1) and seasonal influenza vaccination and disease among adults during the 2009-2010 influenza season. Influenza Other Respir Viruses. 2013 May;7(3):383-92. doi: 10.1111/j.1750-2659.2012.00374.x. Epub 2012 May 9. PMID 22568588
- [Background] Arda B, Durusoy R, Yamazhan T, Sipahi OR, Tasbakan M, Pullukcu H, Erdem E, Ulusoy S. Did the pandemic have an impact on influenza vaccination attitude? A survey among health care workers. BMC Infect Dis. 2011 Apr 7;11:87. doi: 10.1186/1471-2334-11-87. PMID 21473763
- [Background] Halperin BA, MacKinnon-Cameron D, McNeil S, Kalil J, Halperin SA. Maintaining the momentum: key factors influencing acceptance of influenza vaccination among pregnant women following the H1N1 pandemic. Hum Vaccin Immunother. 2014;10(12):3629-41. doi: 10.4161/21645515.2014.980684. PMID 25668670
- [Background] Quinn SC, Parmer J, Freimuth VS, Hilyard KM, Musa D, Kim KH. Exploring communication, trust in government, and vaccination intention later in the 2009 H1N1 pandemic: results of a national survey. Biosecur Bioterror. 2013 Jun;11(2):96-106. doi: 10.1089/bsp.2012.0048. Epub 2013 Apr 25. PMID 23617721
- [Background] Meyer AF, Borkovskiy NL, Brickley JL, Chaudhry R, Franqueira A, Furst JW, Hinsch DM, McDonah MR, Myers JF, Petersen RE, Finney Rutten LJ, Wilson PM, Jacobson RM. Impact of Electronic Point-of-Care Prompts on Human Papillomavirus Vaccine Uptake in Retail Clinics. Am J Prev Med. 2018 Dec;55(6):822-829. doi: 10.1016/j.amepre.2018.06.027. Epub 2018 Oct 19. PMID 30344033
- [Background] Henrikson NB, Zhu W, Baba L, Nguyen M, Berthoud H, Gundersen G, Hofstetter AM. Outreach and Reminders to Improve Human Papillomavirus Vaccination in an Integrated Primary Care System. Clin Pediatr (Phila). 2018 Nov;57(13):1523-1531. doi: 10.1177/0009922818787868. Epub 2018 Jul 13. PMID 30003794
- [Background] Larson HJ, Clarke RM, Jarrett C, Eckersberger E, Levine Z, Schulz WS, Paterson P. Measuring trust in vaccination: A systematic review. Hum Vaccin Immunother. 2018 Jul 3;14(7):1599-1609. doi: 10.1080/21645515.2018.1459252. Epub 2018 May 10. PMID 29617183
- [Background] Karafillakis E, Simas C, Jarrett C, Verger P, Peretti-Watel P, Dib F, De Angelis S, Takacs J, Ali KA, Pastore Celentano L, Larson H. HPV vaccination in a context of public mistrust and uncertainty: a systematic literature review of determinants of HPV vaccine hesitancy in Europe. Hum Vaccin Immunother. 2019;15(7-8):1615-1627. doi: 10.1080/21645515.2018.1564436. Epub 2019 Feb 20. PMID 30633623
- [Background] Holman DM, Benard V, Roland KB, Watson M, Liddon N, Stokley S. Barriers to human papillomavirus vaccination among US adolescents: a systematic review of the literature. JAMA Pediatr. 2014 Jan;168(1):76-82. doi: 10.1001/jamapediatrics.2013.2752. PMID 24276343
- [Background] Fu LY, Bonhomme LA, Cooper SC, Joseph JG, Zimet GD. Educational interventions to increase HPV vaccination acceptance: a systematic review. Vaccine. 2014 Apr 7;32(17):1901-20. doi: 10.1016/j.vaccine.2014.01.091. Epub 2014 Feb 14. PMID 24530401
- [Background] Succi RCM. Vaccine refusal - what we need to know. J Pediatr (Rio J). 2018 Nov-Dec;94(6):574-581. doi: 10.1016/j.jped.2018.01.008. Epub 2018 Apr 12. PMID 29654748
- [Background] Saxena K, Marden JR, Carias C, Bhatti A, Patterson-Lomba O, Gomez-Lievano A, Yao L, Chen YT. Impact of the COVID-19 pandemic on adolescent vaccinations: projected time to reverse deficits in routine adolescent vaccination in the United States. Curr Med Res Opin. 2021 Dec;37(12):2077-2087. doi: 10.1080/03007995.2021.1981842. Epub 2021 Oct 4. PMID 34538163
- [Background] Ryan G, Gilbert PA, Ashida S, Charlton ME, Scherer A, Askelson NM. Challenges to Adolescent HPV Vaccination and Implementation of Evidence-Based Interventions to Promote Vaccine Uptake During the COVID-19 Pandemic: "HPV Is Probably Not at the Top of Our List". Prev Chronic Dis. 2022 Mar 31;19:E15. doi: 10.5888/pcd19.210378. PMID 35358035
- [Background] Patel Murthy B, Zell E, Kirtland K, Jones-Jack N, Harris L, Sprague C, Schultz J, Le Q, Bramer CA, Kuramoto S, Cheng I, Woinarowicz M, Robison S, McHugh A, Schauer S, Gibbs-Scharf L. Impact of the COVID-19 Pandemic on Administration of Selected Routine Childhood and Adolescent Vaccinations - 10 U.S. Jurisdictions, March-September 2020. MMWR Morb Mortal Wkly Rep. 2021 Jun 11;70(23):840-845. doi: 10.15585/mmwr.mm7023a2. PMID 34111058
- [Background] Santoli JM, Lindley MC, DeSilva MB, Kharbanda EO, Daley MF, Galloway L, Gee J, Glover M, Herring B, Kang Y, Lucas P, Noblit C, Tropper J, Vogt T, Weintraub E. Effects of the COVID-19 Pandemic on Routine Pediatric Vaccine Ordering and Administration - United States, 2020. MMWR Morb Mortal Wkly Rep. 2020 May 15;69(19):591-593. doi: 10.15585/mmwr.mm6919e2. PMID 32407298
- [Background] Ateev Mehrotra et al., The Impact of COVID-19 on Outpatient Visits in 2020: Visits Remained Stable, Despite a Late Surge in Cases (Commonwealth Fund, Feb. 2021)
- [Background] Centers for Disease Control and Prevention. Coronavirus Disease 2019 (COVID-19). For Healthcare Professionals. Preserve Supplies. https://www.cdc.gov/coronavirus/2019-ncov/hcp/index.html?CDC_AA_refVal=https%3A%2F%2Fwww.cdc.gov%2Fcoronavirus%2F2019-ncov%2Fhealthcare-facilities%2Findex.html
- [Background] Mann S, Christini K, Chai Y, Chang CP, Hashibe M, Kepka D. Vaccine hesitancy and COVID-19 immunization among rural young adults. Prev Med Rep. 2022 Aug;28:101845. doi: 10.1016/j.pmedr.2022.101845. Epub 2022 Jun 2. PMID 35669235
- [Background] Bar-On YM, Flamholz A, Phillips R, Milo R. SARS-CoV-2 (COVID-19) by the numbers. Elife. 2020 Apr 2;9:e57309. doi: 10.7554/eLife.57309. PMID 32228860
- [Background] Piltch-Loeb R, Silver DR, Kim Y, Norris H, McNeill E, Abramson DM. Determinants of the COVID-19 vaccine hesitancy spectrum. PLoS One. 2022 Jun 1;17(6):e0267734. doi: 10.1371/journal.pone.0267734. eCollection 2022. PMID 35648748
- [Background] Williams CL, Walker TY, Elam-Evans LD, Yankey D, Fredua B, Saraiya M, Stokley S. Factors associated with not receiving HPV vaccine among adolescents by metropolitan statistical area status, United States, National Immunization Survey-Teen, 2016-2017. Hum Vaccin Immunother. 2020 Mar 3;16(3):562-572. doi: 10.1080/21645515.2019.1670036. Epub 2019 Oct 25. PMID 31584312
- [Background] Uva JL, Wagner VL, Gesten FC. Emergency department reliance among rural children in Medicaid in New York State. J Rural Health. 2012 Spring;28(2):152-61. doi: 10.1111/j.1748-0361.2011.00377.x. Epub 2011 Apr 27. PMID 22458316
- [Background] DeGuzman PB, Huang G, Lyons G, Snitzer J, Keim-Malpass J. Rural Disparities in Early Childhood Well Child Visit Attendance. J Pediatr Nurs. 2021 May-Jun;58:76-81. doi: 10.1016/j.pedn.2020.12.005. Epub 2020 Dec 25. PMID 33370620
- [Background] Zablotsky B, Black LI. Prevalence of Children Aged 3-17 Years With Developmental Disabilities, by Urbanicity: United States, 2015-2018. Natl Health Stat Report. 2020 Feb;(139):1-7. PMID 32510313
- [Background] Walker TY, Elam-Evans LD, Yankey D, Markowitz LE, Williams CL, Fredua B, Singleton JA, Stokley S. National, Regional, State, and Selected Local Area Vaccination Coverage Among Adolescents Aged 13-17 Years - United States, 2018. MMWR Morb Mortal Wkly Rep. 2019 Aug 23;68(33):718-723. doi: 10.15585/mmwr.mm6833a2. PMID 31437143
- [Background] Glenn BA, Tsui J, Coronado GD, Fernandez ME, Savas LS, Taylor VM, Bastani R. Understanding HPV vaccination among Latino adolescent girls in three U.S. regions. J Immigr Minor Health. 2015 Feb;17(1):96-103. doi: 10.1007/s10903-014-9996-8. PMID 24557745
- [Background] Mohammed KA, Subramaniam DS, Geneus CJ, Henderson ER, Dean CA, Subramaniam DP, Burroughs TE. Rural-urban differences in human papillomavirus knowledge and awareness among US adults. Prev Med. 2018 Apr;109:39-43. doi: 10.1016/j.ypmed.2018.01.016. Epub 2018 Jan 31. PMID 29378268
- [Background] Shell R, Tudiver F. Barriers to cancer screening by rural Appalachian primary care providers. J Rural Health. 2004 Fall;20(4):368-73. doi: 10.1111/j.1748-0361.2004.tb00051.x. PMID 15551854
- [Background] Peterson CE, Silva A, Holt HK, Balanean A, Goben AH, Dykens JA. Barriers and facilitators to HPV vaccine uptake among US rural populations: a scoping review. Cancer Causes Control. 2020 Sep;31(9):801-814. doi: 10.1007/s10552-020-01323-y. Epub 2020 Jun 14. PMID 32537702
- [Background] Casey MM, Thiede Call K, Klingner JM. Are rural residents less likely to obtain recommended preventive healthcare services? Am J Prev Med. 2001 Oct;21(3):182-8. doi: 10.1016/s0749-3797(01)00349-x. PMID 11567838
- [Background] Yabroff KR, Lawrence WF, King JC, Mangan P, Washington KS, Yi B, Kerner JF, Mandelblatt JS. Geographic disparities in cervical cancer mortality: what are the roles of risk factor prevalence, screening, and use of recommended treatment? J Rural Health. 2005 Spring;21(2):149-57. doi: 10.1111/j.1748-0361.2005.tb00075.x. PMID 15859052
- [Background] Koopman RJ, Mainous AG 3rd, Geesey ME. Rural residence and Hispanic ethnicity: doubly disadvantaged for diabetes? J Rural Health. 2006 Winter;22(1):63-8. doi: 10.1111/j.1748-0361.2006.00009.x. PMID 16441338
- [Background] United States Department of Agriculture. Rural America At a Glance: 2018 Edition. Economic Research Service. Economic Information Bulletin 200. November 2018.
- [Background] Newcomer SR, Freeman RE, Albers AN, Murgel S, Thaker J, Rechlin A, Wehner BK. Missed opportunities for human papillomavirus vaccine series initiation in a large, rural U.S. state. Hum Vaccin Immunother. 2022 Jan 31;18(1):2016304. doi: 10.1080/21645515.2021.2016304. Epub 2022 Feb 4. PMID 35119342
- [Background] Centers for Disease Control and Prevention. Human Papillomavirus (HPV). Cancers Caused by HPV. . Available from: https://www.cdc.gov/hpv/parents/cancer.html
- [Background] Kepka D, Spigarelli MG, Warner EL, Yoneoka Y, McConnell N, Balch A. Statewide analysis of missed opportunities for human papillomavirus vaccination using vaccine registry data. Papillomavirus Res. 2016 Dec;2:128-132. doi: 10.1016/j.pvr.2016.06.002. PMID 27540595
- [Background] Centers for Disease Control and Prevention. HPV-Associated Cancers Rates by Race and Ethnicity. 2019. Atlanta
- [Background] Bruno DM, Wilson TE, Gany F, Aragones A. Identifying human papillomavirus vaccination practices among primary care providers of minority, low-income and immigrant patient populations. Vaccine. 2014 Jul 16;32(33):4149-54. doi: 10.1016/j.vaccine.2014.05.058. Epub 2014 Jun 2. PMID 24886959
- [Background] Katz ML, Reiter PL, Heaner S, Ruffin MT, Post DM, Paskett ED. Acceptance of the HPV vaccine among women, parents, community leaders, and healthcare providers in Ohio Appalachia. Vaccine. 2009 Jun 19;27(30):3945-52. doi: 10.1016/j.vaccine.2009.04.040. Epub 2009 May 3. PMID 19389447
- [Background] Vanderpool RC, Dressler EV, Stradtman LR, Crosby RA. Fatalistic beliefs and completion of the HPV vaccination series among a sample of young Appalachian Kentucky women. J Rural Health. 2015 Spring;31(2):199-205. doi: 10.1111/jrh.12102. Epub 2015 Jan 14. PMID 25640763
- [Background] Blumling AA, Thomas TL, Stephens DP. Researching and Respecting the Intricacies of Isolated Communities. Online J Rural Nurs Health Care. 2013;13(2):Blumling. PMID 24817833
- [Background] Head KJ, Vanderpool RC, Mills LA. Health care providers' perspectives on low HPV vaccine uptake and adherence in Appalachian Kentucky. Public Health Nurs. 2013 Jul;30(4):351-60. doi: 10.1111/phn.12044. Epub 2013 Apr 8. PMID 23808860
- [Background] Henley SJ, Anderson RN, Thomas CC, Massetti GM, Peaker B, Richardson LC. Invasive Cancer Incidence, 2004-2013, and Deaths, 2006-2015, in Nonmetropolitan and Metropolitan Counties - United States. MMWR Surveill Summ. 2017 Jul 7;66(14):1-13. doi: 10.15585/mmwr.ss6614a1. PMID 28683054
- [Background] Centers for Disease Control and Prevention. TeenVaxView. Vaccination Coverage among Adolescents (13 - 17 Years). . Available from: https://www.cdc.gov/vaccines/imz-managers/coverage/teenvaxview/data-reports/index.html
- [Background] U.S. Department of Health and Human Services. Office of Disease Prevention and Health Promotion. Healthy People 2030. Increase the proportion of adolescents who get recommended doses of the HPV vaccine - IID-08. Available from: https://health.gov/healthypeople/objectives-and-data/browse-objectives/vaccination/increase-proportion-adolescents-who-get-recommended-doses-hpv-vaccine-iid-08.
- [Background] Centers for Disease Control and Prevention. How Many Cancers Are Linked with HPV Each Year? Available from: https://www.cdc.gov/cancer/hpv/statistics/cases.htm.
- See also: PREVENT HPV Cancers study website hosted by Kaiser Permanente — https://preventhpvcancers.com/
- See also: PREVENT HPV Cancers study website hosted by Kaiser Permanente — https://research.kpchr.org/preventhpvcancers